CLINICAL TRIAL: NCT05075200
Title: Tranexamic Acid Dosing for Major Joint Replacement Surgery
Acronym: TXA-Dosing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1567
Record Dates: First submitted 2021-09-03; First posted 2021-10-12 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-02

CONDITIONS: Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip
Keywords: Total Knee Arthroplasty; Total Hip Arthroplasty; Tranexamic Acid; TXA; Pharmacokinetics; Dosing; Anti-fibrinolytic
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The main objective of this prospective observational study is to assess TXA blood concentrations in patients requiring major arthroplasty surgery with varied preoperative renal function. We will use this information to create new dosing guidelines for patients undergoing major arthroplasty surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Participants with glomerular filtration rate (GFR) < 60 mL/min/1.73m2 (and dialysis)
  Interventions: Drug: Tranexamic acid
- Group II (Experimental): Participants with GFR ≥ 60 mL/min/1.73m2
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Participants in both groups will be given single intravenous bolus of TXA 20 mg/kg over 15 min after induction of spinal (or other regional technique) or general anesthesia as per standard of care.
  Other Names: CYKLOKAPRON; trans-4 (aminomethyl) cyclohexanecarboxylic acid

SUMMARY:
Over 1.7 million hip and knee replacements are performed every year worldwide. These surgeries are associated with high blood loss and transfusion rates. In older patients, the high blood loss can result in postoperative anemia. Anemia is a condition where there is a lack of healthy red blood cells to carry oxygen around the body. This means, the patient may need a blood transfusion. This can result in different immune responses such as lung injury, fluid overload, and sepsis.

The purpose of this study is to find an optimal dose of tranexamic acid (TXA) to be given during a hip or knee replacement surgery. TXA is one of the drugs given during surgery because it lowers the amount of bleeding and the risk of a blood transfusion.

Individuals who are chosen to participate in the study will be split into two separate groups. After anesthesia is administered, study participant will be given the hospitals standard dose of TXA which is 20mg/kg. However, in patients with kidney problems and lower kidney functions, the dose will be lowered because TXA is filtered out of the body through the kidneys. Throughout the surgery and after it, patients will have about 30-50mL (3-5 tablespoons) of blood samples drawn at specific time points. This will be done through IV line which will stay in place during the surgery and post operation to minimize the amount of needle puncturing's.

This study will help to development a new dosing guideline for TXA in patients who are undergoing joint replacement surgery.

DETAILED DESCRIPTION:
Our study follows a prospective cohort study design without randomization or blinding. 20 patients undergoing unilateral hip or knee replacement will be recruited and stratified into 2 groups (each with 10 patients) with either glomerular filtration rate (GFR) < 60 mL/min/1.73m2 (and dialysis) or GFR ≥ 60 mL/min/1.73m2. This GFR cut-off was chosen based on previous data showing low variability at GFR below and above 60, and plasma TXA levels differed due to reduction in TXA clearance rates between patients in each group.

After spinal/regional or general anesthesia, a single intravenous bolus of 20 mg/kg TXA will be administered (as per our standard of care) over 15 minutes. Serial 4-5 ml blood samples will be drawn at: baseline/pre-TXA administration, 5 min, 15 min, 30 min, 1h, 1.5h, 2h, 6h+/-2h and 12h+/-4h post-bolus. These time points capture 2-3 TXA half-lives, including peak and end of surgery (average 2 h) concentrations.

Each blood sample will be collected into standard citrate collection tubes. Tubes will be inverted a minimum of 5 times to ensure proper mixing with anti-coagulant (sodium citrate). Each sample will be labeled with an anonymized patient study number (to de-identify patient information) and sample time. The tubes will be stored on ice bath following sample collection and then centrifuged within 2 hours at 2000g for about 15 min at 4˚C. The subsequent supernatant will be frozen and stored at -70˚C until analyzed. Measurement of TXA and other drug concentrations, renal biomarkers and metabolomics will be performed using liquid chromatography-tandem mass spectroscopy (LC-MS/MS) using previously described methodology. Patients will otherwise receive routine perioperative care. Patient follow up will be to hospital discharge.

ELIGIBILITY:
Inclusion Criteria

1. Adults > 18 years of age
2. Elective unilateral hip or knee joint replacement

Exclusion Criteria

1. Contraindication to TXA (e.g., allergy, thrombophilia, tretinoin)
2. Advanced liver disease (>2-fold rise in liver enzymes, as this may alter PK analysis)
3. Anti-coagulant use within the last 1-4 days prior (depends on anticoagulant, prior to the day of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jerath, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participants data collected during this trial that underlie the results reported in the publication(s) will be available upon request after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon request immediately after publication of the primary results. No end date.
Access Criteria: Direct request to PI. Anyone who wishes to access the data.

REFERENCES:
- [Derived] Yang Q, He J, Peng HB, Wen B, Idestrup C, Ravi B, Murnaghan J, McCarron A, Hadley H, Shin H, Kaustov L, Wong J, Lin Y, Choi S, Orser BA, Van Der Vyver M, Safa B, Pang KS, Jerath A. Tranexamic Dosing for Major Joint Arthroplasty in Adult Patients with Chronic Kidney Disease: A Pharmacokinetic Study and New Dosing Regimen. Anesthesiology. 2025 May 1;142(5):863-873. doi: 10.1097/ALN.0000000000005397. Epub 2025 Jan 29. PMID 39878614

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I | Group II
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77 [72 to 79] | 72 [63 to 74] | 73 [71 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 7 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 11 | 21
Weight [Median (Inter-Quartile Range); unit: Kilograms] | 80.4 [71.7 to 85.6] | 81 [73 to 112.2] | 81 [71.7 to 101.8]
eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73 m^2] | 46 [42 to 52] | 79 [73 to 83] | 60 [48 to 79]
Surgery type [Count of Participants; unit: Participants]
  Hip Replacement | 4 | 3 | 7
  Knee Replacement | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Blood Plasma TXA Concentration - Total Body Clearance
Description: Measurement of serial blood plasma TXA concentration to build a pharmacokinetic model and dosing regimens for patients within both groups. Curve-stripping of the plasma TXA concentration data according to the 2-compartment model was used to calculate a single value for the measure per participant, which was then averaged.
Time Frame: Collected at 5/15/30/60/90/180/360/540 minutes after bolus
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
mL/min | 58.0 (21.0) | 116 (23.9)

2. Secondary Outcome: Intraoperative Blood Loss and Transfusion
Description: intraoperative measurement of blood loss
Time Frame: Assessed intraoperatively on the day of surgery
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
mL | 100 [100 to 187.5] | 100 [100 to 250]

3. Secondary Outcome: % Change in Pre- and Postoperative Hemoglobin
Description: perioperative value of hemoglobin. The % change is calculated as the postoperative hemoglobin minus preoperative hemoglobin, and reported as a percentage of pre-operative hemoglobin. Negative values indicate a reduction in hemoglobin.
Time Frame: Perioperative
Measure: Mean (Standard Deviation); unit: % decrease
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
% decrease | -14.4 (6.7) | -15.1 (7.9)

4. Secondary Outcome: Postoperative Creatinine
Description: postoperative value of creatinine
Time Frame: Collected within 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
umol/L | 100 [87.25 to 120.75] | 82 [65.5 to 83]

5. Secondary Outcome: Postoperative eGFR
Description: postoperative value of the estimated glomerular filtration rate
Time Frame: Collected within 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: ml/min/1.72 m^2
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
ml/min/1.72 m^2 | 51 [47 to 58] | 85 [78 to 89]

6. Secondary Outcome: In-hospital Mortality
Description: death occurring during the hospital stay
Time Frame: Baseline until hospital discharge (up to 7 days after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

7. Secondary Outcome: Hospital Length of Stay
Description: duration of hospitalization
Time Frame: Baseline until hospital discharge (up to 7 days after surgery)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
hours | 33.2 [30.8 to 57.0] | 29.6 [28.1 to 30.9]

8. Primary Outcome: Blood Plasma TXA Concentration - Area Under the Concentration-time Curve
Description: as for outcome 1
Time Frame: Collected at 5/15/30/60/90/180/360/540 minutes after bolus
Measure: Mean (Standard Deviation); unit: (mg/L)h
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
(mg/L)h | 31031 (10142) | 15808 (3475)

9. Primary Outcome: Blood Plasma TXA Concentration - Elimination Rate Constant
Description: as for outcome 1
Time Frame: Collected at 5/15/30/60/90/180/360/540 minutes after bolus
Measure: Mean (Standard Deviation); unit: /min
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
/min | 0.004 (0.002) | 0.007 (0.002)

10. Primary Outcome: Blood Plasma TXA Concentration - Volume of Central Compartment
Description: as for outcome 1
Time Frame: Collected at 5/15/30/60/90/180/360/540 minutes after bolus
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
L | 13.8 (3.8) | 15.9 (3.2)

11. Primary Outcome: Blood Plasma TXA Concentration - Steady State Volume of Distribution
Description: as for outcome 1
Time Frame: Collected at 5/15/30/60/90/180/360/540 minutes after bolus
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Group I | Group II
Number analyzed (Participants) | 10 | 11
L | 20.9 (6.43) | 25.4 (5.8)

ADVERSE EVENTS:
Time Frame: Baseline until hospital discharge (up to 7 days after surgery)
Arm/Group | Group I | Group II
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT05075200/Prot_SAP_000.pdf